CLINICAL TRIAL: NCT00379340
Title: Treatment of Newly Diagnosed Higher Risk Favorable Histology Wilms Tumors
Brief Title: Combination Chemotherapy With or Without Radiation Therapy in Treating Young Patients With Newly Diagnosed Stage III or Stage IV Wilms' Tumor
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AREN0533; NCI-2009-00419 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AREN0533; CDR0000496508; AREN0533 (Other: Children's Oncology Group); AREN0533 (Other: CTEP); U10CA180886 (NIH); U10CA098543 (NIH)
Record Dates: First submitted 2006-09-19; First posted 2006-09-21 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Stage III Kidney Wilms Tumor; Stage IV Kidney Wilms Tumor
MeSH Terms: conditions — Wilms Tumor | interventions — Radiotherapy, Conformal; Cyclophosphamide; Dactinomycin; Doxorubicin; Etoposide; Vincristine

ARMS (1):
- Treatment (chemotherapy, surgery, radiotherapy) (Experimental): REGIMEN DD4A (weeks 1-6): Patients receive dactinomycin IV; vincristine IV; and doxorubicin hydrochloride IV. Patients with pulmonary and extra-pulmonary metastases at diagnosis undergo radiotherapy.
  Patients with initially unresectable or incompletely resected tumors are reevaluated at week 6, and if resectable, undergo surgery and then proceed to either regimen DD4A or regimen M.
  REGIMEN DD4A (weeks 7-25): Patients receive dactinomycin IV; vincristine IV; and doxorubicin hydrochloride IV.
  REGIMEN M (weeks 7-31): Patients receive cyclophosphamide IV; vincristine IV; and dactinomycin IV and doxorubicin hydrochloride IV. Patients with pulmonary metastases only who are SIR also undergo whole lung radiotherapy.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Procedure: Conventional Surgery; Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Drug: Vincristine Sulfate Liposome

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy
  Other Names: 3-dimensional radiation therapy; 3D Conformal; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D radiotherapy; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy; Radiation, 3D Conformal; Three dimensional external beam radiation therapy (procedure)
Procedure: Conventional Surgery
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Biological: Dactinomycin — Given IV
  Other Names: Actinomycin A IV; Actinomycin C1; Actinomycin D; Actinomycin I1; Actinomycin IV; Actinomycin X 1; Actinomycin-[thr-val-pro-sar-meval]; Cosmegen; DACT; Dactinomycine; Lyovac Cosmegen; Meractinomycin
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
Drug: Vincristine Sulfate Liposome — Given IV
  Other Names: Marqibo

SUMMARY:
This phase III trial is studying how well combination chemotherapy with or without radiation therapy works in treating young patients with newly diagnosed stage III or stage IV Wilms' tumor. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving more than one drug (combination chemotherapy) with or without radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the 4-year event-free survival (EFS) of patients with stage IV favorable histology (FH) Wilms' tumor with pulmonary metastases only who have complete resolution of pulmonary lesions without whole lung irradiation treated with DD4A chemotherapy comprising vincristine, dactinomycin, and doxorubicin hydrochloride.

II. Determine the 4-year EFS of these patients who do not have resolution of pulmonary metastases by week 6 treated with the addition of cyclophosphamide and etoposide to a modified-regimen DD4A (regimen M).

III. Determine the 4-year EFS of patients with stage III or IV FH Wilms' tumor with loss of heterozygosity for chromosomes 1p and 16q treated with regimen M.

SECONDARY OBJECTIVES:

I. Correlate the burden of pulmonary metastatic disease with outcome in patients with stage IV FH Wilms' tumor.

OUTLINE: This is a multicenter study.

REGIMEN DD4A (weeks 1-6): Patients receive dactinomycin IV over 1-5 minutes once in week 1; vincristine IV once in weeks 1-6; and doxorubicin hydrochloride IV over 15 minutes once in week 4 in the absence of disease progression or unacceptable toxicity. Patients with pulmonary and extra-pulmonary metastases at diagnosis undergo radiotherapy once daily beginning in week 1 and continuing for 5-14 days. After completion of DD4A chemotherapy (week 6), patients undergo evaluation. Patients with stage IV disease and pulmonary metastases only with no loss of heterozygosity (LOH) who are rapid complete responders (RCR) (i.e., pulmonary metastases disappear) proceed to regimen DD4A (weeks 7-25).

All other patients (i.e., patients with stage III or IV disease and LOH of both 1p and 16q; stage IV disease with pulmonary metastases only who are slow incomplete responders [SIR] [i.e., pulmonary metastases do not disappear]; or stage IV disease with nonpulmonary metastases or with nonpulmonary metastases in combination with pulmonary metastases) proceed to regimen M (weeks 7-31).

Patients with initially unresectable or incompletely resected tumors are reevaluated at week 6, and if resectable, undergo surgery and then proceed to either regimen DD4A or regimen M as described above.

REGIMEN DD4A (weeks 7-25): Patients receive dactinomycin IV over 1-5 minutes once in weeks 7, 13, 19, and 25; vincristine IV once in weeks 7-10, 13, 16, 19, 22, and 25; and doxorubicin hydrochloride IV over 15 minutes once in weeks 10, 16, and 22 in the absence of disease progression or unacceptable toxicity.

REGIMEN M (weeks 7-31): Patients receive cyclophosphamide IV over 1 hour and etoposide IV over 1 hour on days 1-5 in weeks 7, 10, 19, and 25; vincristine IV once in weeks 8, 9, 11, 12, 13, 16, 22, 28, and 31; and dactinomycin IV and doxorubicin hydrochloride IV over 15 minutes once in weeks 13, 16, 22, 28, and 31 in the absence of disease progression or unacceptable toxicity. Patients with pulmonary metastases only who are SIR also undergo whole lung radiotherapy once daily beginning in week 7 and continuing for 5-14 days.

NOTE: Patients who begin study treatment after undergoing resection of pulmonary metastases are treated according to regimen DD4A (weeks 1-25) and undergo whole lung radiotherapy for 5-14 days beginning in week 1.

After completion of study treatment, patients are followed periodically for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed Wilms' tumor meeting 1 of the following criteria:

  * Stage IV disease with favorable histology with or without loss of heterozygosity (LOH) for 1p and 16q
  * Stage III disease with favorable histology with LOH for 1p and 16q transferring from clinical trial COG-AREN0532
* Patients must begin therapy within 14 days after surgery or biopsy, unless medically contraindicated
* No bilateral Wilms' tumors (stage IV)

  * Patients should be referred to COG-AREN0534
* Previously enrolled in clinical trial COG-AREN03B2
* Karnofsky performance status (PS) 50-100% (for patients > 16 years of age) OR Lansky PS 50-100% (for patients ≤ 16 years of age)
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST or ALT < 2.5 times ULN
* Shortening fraction ≥ 27% by echocardiogram OR ejection fraction ≥ 50% by radionuclide angiogram
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior tumor-directed chemotherapy or radiotherapy unless transferring from clinical trial COG-AREN0532 OR treatment for emergent issues, as medically indicated
* No concurrent aprepitant

Max Age: 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 395 (Actual)
Dates: Start 2007-02-26 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2026-03-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David B Dix, Principal Investigator — Children's Oncology Group
Locations (227):
- United States (199):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Brooklyn Hospital Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Oncology Group, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Cabell-Huntington Hospital, Huntington, West Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (8):
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Children's Hospital-Brisbane, Herston, Queensland
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (16):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Victoria Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- Schneider Children's Medical Center of Israel, Petah Tikua, Israel
- Starship Children's Hospital, Grafton, Auckland, New Zealand
- San Jorge Children's Hospital, San Juan, Puerto Rico
- Swiss Pediatric Oncology Group - Bern, Bern, Switzerland

REFERENCES:
- [Derived] Benedetti DJ, Varela CR, Renfro LA, Tornwall B, Dix DB, Ehrlich PF, Glick RD, Kalapurakal J, Perlman E, Gratias E, Seibel NL, Geller JI, Khanna G, Malogolowkin M, Grundy P, Fernandez CV, Dome JS, Mullen EA. Treatment of children with favorable histology Wilms tumor with extrapulmonary metastases: A report from the COG studies AREN0533 and AREN03B2 and NWTSG study NWTS-5. Cancer. 2024 Mar 15;130(6):947-961. doi: 10.1002/cncr.35099. Epub 2023 Nov 7. PMID 37933882
- [Derived] Madanat-Harjuoja LM, Renfro LA, Klega K, Tornwall B, Thorner AR, Nag A, Dix D, Dome JS, Diller LR, Fernandez CV, Mullen EA, Crompton BD. Circulating Tumor DNA as a Biomarker in Patients With Stage III and IV Wilms Tumor: Analysis From a Children's Oncology Group Trial, AREN0533. J Clin Oncol. 2022 Sep 10;40(26):3047-3056. doi: 10.1200/JCO.22.00098. Epub 2022 May 17. PMID 35580298
- [Derived] Dix DB, Fernandez CV, Chi YY, Mullen EA, Geller JI, Gratias EJ, Khanna G, Kalapurakal JA, Perlman EJ, Seibel NL, Ehrlich PF, Malogolowkin M, Anderson J, Gastier-Foster J, Shamberger RC, Kim Y, Grundy PE, Dome JS; AREN0532 and AREN0533 study committees. Augmentation of Therapy for Combined Loss of Heterozygosity 1p and 16q in Favorable Histology Wilms Tumor: A Children's Oncology Group AREN0532 and AREN0533 Study Report. J Clin Oncol. 2019 Oct 20;37(30):2769-2777. doi: 10.1200/JCO.18.01972. Epub 2019 Aug 26. PMID 31449468
- [Derived] Dix DB, Seibel NL, Chi YY, Khanna G, Gratias E, Anderson JR, Mullen EA, Geller JI, Kalapurakal JA, Paulino AC, Perlman EJ, Ehrlich PF, Malogolowkin M, Gastier-Foster JM, Wagner E, Grundy PE, Fernandez CV, Dome JS. Treatment of Stage IV Favorable Histology Wilms Tumor With Lung Metastases: A Report From the Children's Oncology Group AREN0533 Study. J Clin Oncol. 2018 Jun 1;36(16):1564-1570. doi: 10.1200/JCO.2017.77.1931. Epub 2018 Apr 16. PMID 29659330
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The 15 discrepant patients were ineligible to the study. They were excluded in the Participant Flow table because none of them were treated by the protocol and their group designations were unknown.
Groups:
- Stage IV and Rapid Complete Response (RCR) of Lung Metastases: Stage IV and rapid complete response (RCR) of lung metastases continuously treated with DD4A after 6 weeks of DD4A.
- Stage IV and Slow Incomplete Response (SIR) of Lung Metastases: Stage IV and slow incomplete response (SIR) of lung metastases treated with Regimen M after 6 weeks of DD4A.
- Stage III/IV With LOH 1p and 16q Treated With Regimen M: Stage III/IV with LOH 1p and 16q treated with Regimen M.
- Stage IV With Non-lung Disease Treated With Regimen M: Stage IV with non-lung disease treated with Regimen M.
- Stage IV With Lung Metastases: Stage IV with lung metastases treated with DD4A for less than 6 weeks and/or response inevaluable at week 6.
Period: Overall Study
Arm/Group | Stage IV and Rapid Complete Response (RCR) of Lung Metastases | Stage IV and Slow Incomplete Response (SIR) of Lung Metastases | Stage III/IV With LOH 1p and 16q Treated With Regimen M | Stage IV With Non-lung Disease Treated With Regimen M | Stage IV With Lung Metastases
Started | 120 | 135 | 52 | 50 | 23
Completed | 107 | 132 | 50 | 37 | 9
Not Completed | 13 | 3 | 2 | 13 | 14
Not completed — Death | 0 | 0 | 0 | 2 | 0
Not completed — Lack of Efficacy | 6 | 1 | 0 | 4 | 3
Not completed — Physician Decision | 6 | 2 | 1 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0
Not completed — Refusal of further protocol therapy | 1 | 0 | 1 | 1 | 7
Not completed — On more than 1 tumor therapeutic study | 0 | 0 | 0 | 2 | 0
Not completed — Delayed nephrectomy and anaplasia | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage IV and Rapid Complete Response (RCR) of Lung Metastases | Stage IV and Slow Incomplete Response (SIR) of Lung Metastases | Stage III/IV With LOH 1p and 16q Treated With Regimen M | Stage IV With Non-lung Disease Treated With Regimen M | Stage IV With Lung Metastases | Total
Number analyzed (Participants) | 120 | 135 | 52 | 50 | 23 | 380
Age, Continuous [Mean (Standard Deviation); unit: Months] | 54.94 (36.27) | 55.07 (27.16) | 52.16 (28.64) | 69.58 (39.24) | 56.06 (23.71) | 56.60 (32.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 71 | 30 | 31 | 8 | 205
  Male | 55 | 64 | 22 | 19 | 15 | 175
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 18 | 6 | 12 | 3 | 51
  Not Hispanic or Latino | 104 | 108 | 42 | 36 | 18 | 308
  Unknown or Not Reported | 4 | 9 | 4 | 2 | 2 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 2 | 2 | 0 | 2 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 21 | 22 | 10 | 4 | 1 | 58
  White | 80 | 94 | 38 | 39 | 18 | 269
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 16 | 17 | 4 | 5 | 3 | 45

OUTCOME MEASURES:

1. Primary Outcome: Event Free Survival Probability
Description: Probability of no relapse, secondary malignancy, or death after 4 year in the study.
Time Frame: 4 years
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Stage IV and Rapid Complete Response (RCR) of Lung Metastases
Number analyzed (Participants) | 120
Probability | 0.79 [0.70 to 0.87]

2. Primary Outcome: Event Free Survival (EFS) Probability
Description: Probability of no relapse, secondary malignancy, or death after 4 year in the study.
Time Frame: At 4 years
Population: Analysis includes only eligible patients.
Measure: Number (95% Confidence Interval); unit: Probability of EFS at 4 years
Groups:
- Stage IV and Slow Incomplete Response (SIR) of Lung Metastases: Stage IV and slow incomplete response (SIR) of lung metastases treated with Regimen M after 6 weeks of DD4A
  doxorubicin hydrochloride: Given IV
  liposomal vincristine sulfate: Given IV
  conventional surgery
  3-dimensional conformal radiation therapy
  dactinomycin: Given IV
  cyclophosphamide: Given IV
  etoposide: Given IV
Arm/Group | Stage IV and Slow Incomplete Response (SIR) of Lung Metastases
Number analyzed (Participants) | 135
Probability of EFS at 4 years | 0.89 [0.82 to 0.95]

3. Primary Outcome: Event Free Survival Probability
Description: Probability of no relapse, secondary malignancy, or death after 4 year in the study
Time Frame: At 4 years
Population: All eligible patients were included in this analysis.
Measure: Number (95% Confidence Interval); unit: Probability of EFS at 4 years
Groups:
- Stage III/IV With LOH 1p and 16q Treated With Regimen M: Stage III/IV with LOH 1p and 16q treated with Regimen M
  doxorubicin hydrochloride: Given IV
  liposomal vincristine sulfate: Given IV
  conventional surgery
  3-dimensional conformal radiation therapy
  dactinomycin: Given IV
  cyclophosphamide: Given IV
  etoposide: Given IV
- Stage IV With Non-lung Disease Treated With Regimen M: Stage IV with non-lung disease treated with Regimen M
  doxorubicin hydrochloride: Given IV
  liposomal vincristine sulfate: Given IV
  conventional surgery
  dactinomycin: Given IV
  cyclophosphamide: Given IV
  etoposide: Given IV
Arm/Group | Stage III/IV With LOH 1p and 16q Treated With Regimen M | Stage IV With Non-lung Disease Treated With Regimen M
Number analyzed (Participants) | 52 | 50
Probability of EFS at 4 years | 0.90 [0.80 to 1] | 0.73 [0.59 to 0.88]

4. Secondary Outcome: Event Free Survival Associated With the Burden of Pulmonary Metastatic Disease
Description: Probability of no relapse, secondary malignancy, or death after 4 year in the study.
Time Frame: At 4 years
Population: Analysis population is eligible stage (stg) IV patients (pts) with lung mets only. On Participant Flow table, these pts include 120 RCR, 135 SIR, 21 stg IV with LOH (of 52 when including stg III), and 23 stg IV with lung mets (off therapy before week 6). A total of 299 stg IV pts, exceeding the total number of participant (297) analyzed for OM 4.
Measure: Number (95% Confidence Interval); unit: Probability
Groups:
- Lung Mets <= 1cm: Lung mets <= 1cm
- Lung Mets > 1cm: Lung mets > 1cm
Arm/Group | Lung Mets <= 1cm | Lung Mets > 1cm
Number analyzed (Participants) | 147 | 150
Probability | 0.88 [0.82 to 0.95] | 0.82 [0.75 to 0.90]

ADVERSE EVENTS:
Arm/Group | Stage IV and Rapid Complete Response (RCR) of Lung Metastases | Stage IV and Slow Incomplete Response (SIR) of Lung Metastases | Stage III/IV With LOH 1p and 16q Treated With Regimen M | Stage IV With Non-lung Disease Treated With Regimen M | Stage IV With Lung Metastases
Serious Adverse Events (participants affected / at risk) | 3/120 | 10/135 | 3/52 | 11/50 | 0/23
Other Adverse Events (participants affected / at risk) | 11/120 | 90/135 | 35/52 | 37/50 | 1/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage IV and Rapid Complete Response (RCR) of Lung Metastases (N=120) | Stage IV and Slow Incomplete Response (SIR) of Lung Metastases (N=135) | Stage III/IV With LOH 1p and 16q Treated With Regimen M (N=52) | Stage IV With Non-lung Disease Treated With Regimen M (N=50) | Stage IV With Lung Metastases (N=23)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CPK increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death NOS (General disorders) | 2 (2) | 3 (3) | 2 (2) | 3 (3) | 0 (0)
Hepatobiliary disorders - Other specify (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign malignant and unspecified (incl cy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory thoracic and mediastinal disorders - Ot (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage IV and Rapid Complete Response (RCR) of Lung Metastases (N=120) | Stage IV and Slow Incomplete Response (SIR) of Lung Metastases (N=135) | Stage III/IV With LOH 1p and 16q Treated With Regimen M (N=52) | Stage IV With Non-lung Disease Treated With Regimen M (N=50) | Stage IV With Lung Metastases (N=23)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 5 (6) | 3 (3) | 6 (6) | 1 (1)
Anaphylaxis (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 3 (4) | 2 (2) | 2 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 10 (12) | 5 (7) | 9 (14) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 1 (1)
Bladder infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood and lymphatic system disorders - Other specif (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 10 (10) | 3 (3) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Duodenal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 53 (77) | 21 (27) | 20 (23) | 1 (2)
Fever (General disorders) | 0 (0) | 5 (6) | 0 (0) | 1 (1) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
GGT increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hepatobiliary disorders - Other specify (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 3 (4) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 3 (5) | 0 (0) | 3 (4) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 3 (3) | 3 (3) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 6 (6) | 6 (6) | 3 (3) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (1) | 3 (4) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Ileal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Infections and infestations - Other specify (Infections and infestations) | 2 (2) | 20 (22) | 11 (17) | 9 (11) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Jejunal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 4 (4) | 2 (2) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 4 (4) | 2 (2) | 3 (3) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 5 (5) | 2 (3) | 4 (4) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 4 (6) | 3 (5) | 2 (2) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 4 (5) | 3 (4) | 2 (5) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 3 (4) | 3 (4) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Soft tissue necrosis lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stoma site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 3 (4) | 2 (3) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3) | 2 (3) | 4 (5) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular disorders - Other specify (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3) | 6 (7) | 1 (1)
Vulval infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (1) | 2 (2) | 3 (4) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 2 (3) | 2 (2) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.